CLINICAL TRIAL: NCT04334811
Title: Stereotactic Ablative Radiotherapy (SAbR) for Treatment of Ventricular Tachycardia (VT) Refractory Standard Invasive Ablation Techniques
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to participation in a multi-center randomized controlled trial with competing enrollment criteria.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James Daniels, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1023
Record Dates: First submitted 2020-02-20; First posted 2020-04-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Tachycardia, Ventricular
Keywords: heart
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Arm (Other): No arm
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — Stereotactic ablative radiotherapy (SAbR) delivers of a potent, ablative or nearly ablative dose of radiation in oligofractions (ie, five or fewer fractions) primarily to create a compact dose delivered accurately to the intended target with steep gradients in all directions (geometric avoidance) and avoid damaging normal tissues.
  Other Names: SAbR

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of stereotactic ablative radiotherapy (SAbR), also known as stereotactic body radiation therapy (SBRT), for treatment of ventricular tachycardia (VT) requiring implantable cardioverter defibrillator (ICD) treatments in patients with VT refractory to standard invasive ablation techniques. We hypothesized that SAbR is effective in suppressing sustained VT and reducing ICD treatments in this group of patients and is associated with acceptably low risk of serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have an ICD implanted > 6 months and all VT episodes in the past 6 months are available in device memory.
* Within the past 3 months, the patient has at least one episode of symptomatic monomorphic VT that requires ICD treatment (anti-tachycardia pacing and/or ICD shock) or was sustained/incessant but falls under ICD treatment zone. These VT episodes must occur after at least one standard invasive VT ablation or occur in a patient that is clinically deemed not eligible to the standard VT ablation procedure.
* Two independent cardiac electrophysiologists reviewed the case and agreed that the patient would benefit from suppression of these VT episodes but there is no optimal invasive VT ablation or antiarrhythmic drug options.

Exclusion Criteria:

* Has contraindication to receive SAbR or VT clinically deemed not suitable for SAbR.
* Is pregnant
* Has severe co-morbid medical condition or terminal illness and is unlikely to survive more than 6 months regardless of VT status based on clinical judgement by treating or enrolling physicians.
* On potent immunosuppressive therapy (e.g., post organ transplant)
* Has severe collagen vascular disorder with organ involvement
* Not willing or not able to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome of ICD (implantable cardioverter-defibrillator) Treatment | 6 months
  Number of episodes of ICD (implantable cardioverter-defibrillator) treatment (including both ATP and shock) per month; comparing 6 months before and after SAbR (excluding the first 2-week blanking period post SAbR).

CONTACTS AND LOCATIONS:
Overall Officials: James Daniel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States